CLINICAL TRIAL: NCT00352157
Title: Effect of Revival Soy on Weight Loss and Appearance of Skin, Hair, and Nails in High BMI Premenopausal Women
Brief Title: Effect of Revival Soy on Weight Loss and Skin, Hair, and Nails in Premenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Physicians Pharmaceuticals, Inc. (Industry)
Collaborators: Dermatology Consulting Services, High Point NC (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DCS-61-06
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2009-07-21 (Estimated); Status verified 2009-07

CONDITIONS: Skin Aging; Weight Loss
Keywords: Soy; Dermatology; Skin; Hair; Finger Nails; Weight Loss; Body Mass Index; Photoaging of Skin; Skin Wrinkling
MeSH Terms: conditions — Weight Loss

INTERVENTIONS:
Behavioral: Revival Soy Dietary Supplement

SUMMARY:
The purpose of this study is to determine if dietary consumption of Revival Soy can improve the appearance of the skin, hair, and finger nails and support weight loss in overweight, premenopausal women.

DETAILED DESCRIPTION:
The researchers hypothesize that supplementation of Revival® Soy products to overweight premenopausal women as part of a soy-based meal replacement diet plan will:

* Improve the health and appearance of the skin by normalizing skin pigmentation and reducing wrinkles,
* Improve the health and appearance of hair by enhancing sheen and ease of combing, and
* Improve the health and appearance of nails by enhancing shine, flexibility, and strength.
* Stimulate a loss in weight and a reduction in the Body Mass Index (BMI),

For this study, obese (BMI = 30-40 kg/m2) premenopausal women (25-45 years of age) with mild to moderate photoaging (n=40) will receive either a Revival® soy shake (20 grams soy protein with 160 mg total isoflavones; n=20) or a placebo shake (20 grams of milk protein with 0 mg isoflavones; n=20) daily for 6 months. The subjects will be asked to come into the office for a total of seven visits, at baseline and at monthly intervals for 6 months. At baseline, month 3, and month 6, the subjects will be asked to complete a questionnaire in order to provide self-reported improvements related to hair, skin, and nail health. Following completion of the questionnaire, the investigator and the dermatology clinic staff will examine the subjects to assess the health and appearance of their skin, hair, and nails at baseline, month 3, and month 6.

After acceptance into the study, a registered dietitian will instruct the study subjects in the use of a low-energy (1,200 - 1,500 kcal/day) diet that incorporates 2 soy-based daily meal replacements (shakes, ~500 kcal), a minimum of 5 daily servings of fruits and vegetables (~300 kcal), and one entrée (~400 - 500 kcal). Subjects will be required to keep a dietary food intake record of all food and supplement use during the trial. Anthropometric data (height, body weight, waist circumference and hip circumference) will be collected at baseline and at monthly intervals.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Age: 25-45 years.
* BMI between 30 - 40 kg/m2.
* Motivated to lose weight.
* Subjects must be in general good health as determined from a medical history.
* Subjects must have mild to moderate photoaging.
* Subjects must use a shampoo from the approved list without change for the entire duration of the study.
* Must not be consuming soy supplements or other soy products currently.
* Must not be pregnant (negative pregnancy test at screening) and agree not to become pregnant during the course of the study.
* Subjects must read and sign the informed consent form after the nature of the study has been fully explained.

Exclusion Criteria:

* Subjects with known allergies or sensitivities to ingredients contained in the dietary supplement.
* Subjects who are required to spend excessive time in the sun (i.e. lifeguards, other outdoor workers).
* Subjects who are currently participating or have participated within the last 4 weeks in any other clinical study (i.e., dermal patch, use tests, investigational drug or devices, etc.).
* Subjects viewed by the investigator as not being able to complete the study.
* Subjects who are unwilling to leave all of their current skin care products unchanged for the 6 months of the study.
* Subjects who are unwilling to leave all of their current nail care products unchanged for the 6 months of the study.
* Subjects who are unwilling to leave all of their current oral medications unchanged for the 6 months of the study.
* Subjects who have experienced large variations in body weight during the previous 3 months
* Subjects currently using other weight loss medications or supplements.
* Subjects who had surgical intervention for the treatment of obesity.

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2006-07; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Investigator assessed appearance of skin (roughness, wrinkling, dyspigmentation, and redness) at baseline and after 3 and 6 months
Investigator assessed appearance of hair (roughness, dullness, lack of manageability, and scalp flaking) at baseline and after 3 and 6 months
Investigator assessed appearance of finger nails (roughness, ridging, flaking, and splitting) at baseline and after 3 and 6 months.

SECONDARY OUTCOMES:
Body weight at monthly intervals
Body mass index (BMI) at the baseline and study completion
Subject-perceived changes in appearance of skin, hair, and finger nails at baseline and after 3 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Zoe D Draelos, M.D., Principal Investigator — Dermatology Consulting Services, High Point NC
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States